CLINICAL TRIAL: NCT04472026
Title: Adequate Selection of Patients for Thyroid Biopsy: Evaluation of a Shared Decision Making Conversation Aid
Brief Title: AIM1: Adequate Selection of Patients for Thyroid Biopsy: Evaluation of a Shared Decision Making Conversation Aid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB202000837; K08CA248972 (NIH)
Record Dates: First submitted 2020-07-10; First posted 2020-07-15 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Thyroid Nodules; Thyroid Cancer
Keywords: thyroid nodules; shared decision making
MeSH Terms: conditions — Thyroid Nodule; Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Counseling using the electronic conversation aid
  Interventions: Behavioral: Counseling using the electronic conversation aid

INTERVENTIONS:
Behavioral: Counseling using the electronic conversation aid — This conversation aid will help you and your doctor discuss ways to care for your thyroid nodule. We will evaluate the acceptability of the conversation aid and barriers to implementation in clinical practice. Post visit semi structured interviews and recordings of the clinical visits will be qualitatively analyzed. We hypothesize that the conversation aid will be accepted and facilitate the decision making process.

SUMMARY:
There is an epidemic of thyroid cancer that is harmful to patients and the medical system. The study hypothesizes that the use of an electronic conversation aid during clinical visits can help patients and clinicians collaborate when deciding the next step in management for a thyroid nodule. The study aims to update a conversation aid prototype that was developed to support shared decision making in the diagnosis of thyroid cancer. This entry (Aim 1) has an associated study (Aim 2) registered under NCT04463719

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years old presenting for evaluation of a thyroid nodule

Exclusion Criteria:

* Patients with hyperthyroidism
* Patients with previous biopsy of the nodule of interest
* Pregnant patients
* Prisoners

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naykky Singh Ospina, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study aims to update a conversation aid prototype that was developed to support shared decision making in the diagnosis of thyroid cancer. Adult patients with thyroid nodules presenting for consultation were recruited from two clinical centers (University of Florida, Gainesville and Mayo Clinic, Rochester). Enrollment started on 07/16/2020 and was completed on 08/02/2021.
Period: Overall Study
Arm/Group | Intervention Group
Started (Patients and clinicians starting the study. Guest are not considered as units of analysis/participants.) | 66
Clinicians Starting | 13 (Clinicians)
Clinicians Completing | 12
Patients Starting | 53
Patient Completing | 49
Completed (Patients and clinicians completing the study) | 61
Not Completed | 5
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Population: Patients and clinicians included in the study and are reported individually and not as dyads. Clinicians age, race/ethnicity were not collected (0 noted below). The patient data is used to describe the overall age of the population. No information was collected from guest.
Groups:
- Intervention Group: Patients: Counseling using the electronic conversation aid
  Counseling using the electronic conversation aid: This conversation aid will help you and your doctor discuss ways to care for your thyroid nodule. We will evaluate the acceptability of the conversation aid and barriers to implementation in clinical practice. Post visit semi structured interviews and recordings of the clinical visits will be qualitatively analyzed. We hypothesize that the conversation aid will be accepted and facilitate the decision making process.
- Intervention Group: Clinicians: Counseling using the electronic conversation aid
  Counseling using the electronic conversation aid: This conversation aid will help you and your patient discuss ways to care for their thyroid nodule. We will evaluate the acceptability of the conversation aid and barriers to implementation in clinical practice. Post visit semi structured interviews and recordings of the clinical visits will be qualitatively analyzed. We hypothesize that the conversation aid will be accepted and facilitate the decision making process.
- Total: Total of all reporting groups
Arm/Group | Intervention Group: Patients | Intervention Group: Clinicians | Total
Number analyzed (Participants) | 53 | 13 | 66
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Age was not collected from clinicians
  years
    number analyzed (Participants) | 53 | 0 | 53
    (all) | 62 [53 to 70] |  | 62 [53 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 8 | 50
  Male | 11 | 5 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity not collected for clinicians.
  Participants
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 53 | 0 | 53
    Unknown or Not Reported | 0 | 13 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race not collected for clinicians.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 5 | 0 | 5
    White | 47 | 0 | 47
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 1 | 13 | 14

OUTCOME MEASURES:

1. Primary Outcome: Qualitative Analysis of the Patient and Clinician Experience Using the Conversation Aid
Description: The clinical visit and post visit semi-structure interviews of patient and clinicians that have used the conversation aid will be analyzed qualitatively to better understand the acceptability of the conversation aid in clinical practice and used to further update the conversation aid.
Time Frame: Up to the time the post visit interview was completed (on average 1 weeks after the clinical visit for patients and 1 month after completion of 3 visit using the tool for clinicians)
Measure: Count of Participants; unit: Participants
Groups:
- Patients Receiving Care With the Conversation Aid: Post visit semi structured interviews and recordings of the clinical visits of patients who received care with the conversation aid
- Clinician Providing Care With the Conversation Aid: Review of clinical visit and post visit interviews of clinicians providing care with the conversation aid
Arm/Group | Patients Receiving Care With the Conversation Aid | Clinician Providing Care With the Conversation Aid
Number analyzed (Participants) | 49 | 12
Participants
  Positive (tool features and components) | 12 | 0
  Positive (Understanding the medical condition, situation and options) | 12 | 0
  Positive (Interaction with the clinician) | 12 | 0
  Negative (Suggestions for improvement related to TNOC features/components) | 7 | 0
  Negative (Impact on the interaction) | 6 | 0
  Positive (tool features) | 0 | 4
  Positive (benefits patients) | 0 | 4
  Positive (benefits clinicians) | 0 | 2
  Negative (using TNOC is a change in their routine) | 0 | 1
  Negative (Improvements to support the use of TNOC in routine Practice) | 0 | 1

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed due to the nature of the intervention.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed due to the nature of the intervention. The intervention in this study was the use of a conversation aid during the clinical visit. No medication, drug, or test were performed during the study.
Arm/Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/26/NCT04472026/Prot_SAP_ICF_000.pdf